CLINICAL TRIAL: NCT04046666
Title: Difference in the Metabolic Characteristics of COPD Patients and Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019ZY005-MERIDIAN
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: meridians; acupuncture; chronic obstructive pulmonary disease; meridian phenomenon; near infrared spectroscopy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Moxibustion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COPD group (Other): This group will include 40 patients with chronic obstructive pulmonary disease (COPD).
  Interventions: Device: Functional near infrared spectroscopy
- Healthy group (Other): This group will include 40 healthy volunteers.
  Interventions: Device: Functional near infrared spectroscopy
- Healthy intervention group (Other): This group will include 40 healthy volunteers, who will receive moxibustion intervention.
  Interventions: Device: Functional near infrared spectroscopy; Procedure: Moxibustion

INTERVENTIONS:
Device: Functional near infrared spectroscopy — Functional near infrared spectroscopy will be adopted to assess the metabolic characteristics of the Heart and Lung meridians. The probes will be left at 4 measurement sites, which include Shenmen (HT7) and Shaohai (HT3) of the Heart meridian, Taiyuan (LU9) and Chize (LU5) of the Lung meridian.
Procedure: Moxibustion — Two sessions of moxibustion will be performed in the Heart meridian and Lung meridian successively.
  Intervention in the Heart meridian: moxibustion will be performed above Shaohai (HT3) for 15 minutes. During moxibustion, the probes of near infrared spectroscopy will detect the metabolic characteristics of three measuring sites, which include the midpoint of the Heart meridian along the forearm, Chize (LU5) of the Lung meridian, and the midpoint of the Lung meridian along the forearm.
  Intervention in the Lung meridian: moxibustion will be performed above Chize (LU5) for 15 minutes. During moxibustion, the probes of near infrared spectroscopy will detect the metabolic characteristics of three measuring sites, which include the midpoint of the Lung meridian along the left forearm, Shaohai (HT3) of the Heart meridian, and the midpoint of the Heart meridian along the forearm.
  Arms: Healthy intervention group

SUMMARY:
Although some important progresses were made in the field of the meridian research, no breakthroughs have been achieved. Besides,there are some problems in meridian researches. Particularly, previous research of meridian phenomenon involved lots of subjective elements and outcomes.Researches that use modern scientific techniques to investigate the biological characteristics of meridians are urgently needed. Therefore, this study is designed to assess the metabolic characteristics of the Heart and Lung meridians by using functional near infrared spectroscopy. Thus, the biological characteristics of meridians could be presented objectively in a scientific methodology.

DETAILED DESCRIPTION:
The Lung and Heart meridians are chosen as two specific studied meridians. Participants of chronic obstructive pulmonary disease (COPD) and healthy volunteers will be enrolled.

120 participants will be included and divided into the healthy control group, chronic obstructive pulmonary disease (COPD) group and healthy intervention group. Functional near infrared spectroscopy will be used to assess the metabolic characteristics of the Heart and Lung meridians. The specificity for the meridian-visceral association will be investigated by comparing the metabolic difference between the Heart and Lung meridians in the healthy control group and COPD group. Besides, participants in the healthy intervention group will receive two sessions of moxibustion in the Heart meridian and Lung meridian respectively to explore the specificity for the site-to-site association.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for COPD

1. Patients should meet the above diagnostic criteria, and the severity of COPD is in the stage of GOLD 2 or 3 based on pulmonary function testing;
2. COPD patients in the stable phase, who present with mild symptoms of cough, expectoration and short breath;
3. 35 ≤ age ≤75 years, male or female;
4. Patients have clear consciousness and could communicate with others normally;
5. Patients could understand the full study protocol and written informed consent is signed by themselves or their lineal kin.

Inclusion criteria for health volunteers

1. Healthy volunteers who could provide a recent medical examination report to confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological disease;
2. Age≥20 years, male or female;
3. Participants have clear consciousness and could communicate with others normally;
4. Participants could understand the full study protocol and have high adherence .Written informed consent is signed by themselves or their lineal kin.

Exclusion Criteria:

Exclusion criteria for COPD

1. Patients who fail to meet the diagnostic criteria for COPD, or COPD patients in the phase of acute exacerbation;
2. Patients have the following complications, which includes pneumonia, bronchial asthma, bronchiectasis, active tuberculosis, pneumothorax, chest trauma, tumors of the lung or thorax, and other confirmed respiratory diseases;
3. Patients have concomitant conditions of heart diseases, such as chronic stable angina pectoris;
4. Patients have serious concomitant conditions and fail to treat them effectively, such as diseases of the digestive, urinary, respiratory, hematological, and nervous system;
5. Patients have mental illness, severe depression, alcohol dependence or history of drug abuse;
6. Pregnant or lactating patients;
7. Patients are participating in other trials.

Exclusion criteria of health volunteers

1. Participants have sudden severe diseases during the trial, such as cardiovascular diseases, liver diseases, kidney diseases, urinary diseases and hematological diseases.
2. Participants have mental illness, severe depression, alcohol dependence or history of drug abuse;
3. Pregnant or lactating participants ;
4. Participants are participating in other trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline regional oxygen saturation (rSO2) | 5-minute baseline, 15 minutes during moxibustion and 5 minutes after removal of moxibustion
  Regional oxygen saturation could reflect the metabolic characteristics of meridians.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litscher G, Wang L. [Cerebral near infrared spectroscopy and acupuncture--results of a pilot study]. Biomed Tech (Berl). 2000 Jul-Aug;45(7-8):215-8. doi: 10.1515/bmte.2000.45.7-8.215. German. PMID 10975151
- [Background] Raith W, Pichler G, Sapetschnig I, Avian A, Sommer C, Baik N, Koestenberger M, Schmolzer GM, Urlesberger B. Near-infrared spectroscopy for objectifying cerebral effects of laser acupuncture in term and preterm neonates. Evid Based Complement Alternat Med. 2013;2013:346852. doi: 10.1155/2013/346852. Epub 2013 May 15. PMID 23762122
- [Background] Litscher G, Wang L, Huber E. [Changes in cerebral near infrared spectroscopy parameters during manual acupuncture needle stimulation]. Biomed Tech (Berl). 2002 Apr;47(4):76-9. doi: 10.1515/bmte.2002.47.4.76. German. PMID 12051136
- [Background] Takamoto K, Hori E, Urakawa S, Sakai S, Ishikawa A, Kohno S, Ono T, Nishijo H. Cerebral hemodynamic responses induced by specific acupuncture sensations during needling at trigger points: a near-infrared spectroscopic study. Brain Topogr. 2010 Sep;23(3):279-91. doi: 10.1007/s10548-010-0148-8. Epub 2010 May 26. PMID 20502956
- [Background] Litscher G, Wang L, Schwarz G, Schikora D. [Increases of intracranial pressure and changes of blood flow velocity due to acupressure, needle and laser needle acupuncture?]. Forsch Komplementarmed Klass Naturheilkd. 2005 Aug;12(4):190-5. doi: 10.1159/000087044. Epub 2005 Aug 29. German. PMID 16137980
- [Background] Litscher G, Schwarz G, Sandner-Kiesling A, Hadolt I, Eger E. Effects of acupuncture on the oxygenation of cerebral tissue. Neurol Res. 1998;20 Suppl 1:S28-32. doi: 10.1080/01616412.1998.11740605. PMID 9584920
- [Background] Ohkubo M, Hamaoka T, Niwayama M, Murase N, Osada T, Kime R, Kurosawa Y, Sakamoto A, Katsumura T. Local increase in trapezius muscle oxygenation during and after acupuncture. Dyn Med. 2009 Mar 16;8:2. doi: 10.1186/1476-5918-8-2. PMID 19291290
- [Background] Litscher G, Ofner M, He W, Wang L, Gaischek I. Acupressure at the Meridian Acupoint Xiyangguan (GB33) Influences Near-Infrared Spectroscopic Parameters (Regional Oxygen Saturation) in Deeper Tissue of the Knee in Healthy Volunteers. Evid Based Complement Alternat Med. 2013;2013:370341. doi: 10.1155/2013/370341. Epub 2013 Feb 7. PMID 23476689
- [Background] Banzer W, Hubscher M, Seib M, Vogt L. Short-time effects of laser needle stimulation on the peripheral microcirculation assessed by laser Doppler spectroscopy and near-infrared spectroscopy. Photomed Laser Surg. 2006 Oct;24(5):575-80. doi: 10.1089/pho.2006.24.575. PMID 17069486
- [Background] Jimbo S, Atsuta Y, Kobayashi T, Matsuno T. Effects of dry needling at tender points for neck pain (Japanese: katakori): near-infrared spectroscopy for monitoring muscular oxygenation of the trapezius. J Orthop Sci. 2008 Mar;13(2):101-6. doi: 10.1007/s00776-007-1209-z. Epub 2008 Apr 8. PMID 18392913
- [Background] Murkin JM, Arango M. Near-infrared spectroscopy as an index of brain and tissue oxygenation. Br J Anaesth. 2009 Dec;103 Suppl 1:i3-13. doi: 10.1093/bja/aep299. PMID 20007987
- [Derived] Jiang Y, Hu H, Li X, He X, Shao X, Lou J, Zhang Y, Wu Y, Fang J. Difference in the metabolic characteristics of chronic obstructive pulmonary disease patients and healthy adults. Medicine (Baltimore). 2020 Jul 24;99(30):e21302. doi: 10.1097/MD.0000000000021302. PMID 32791715